CLINICAL TRIAL: NCT04274361
Title: Ketamine Infusion for Pain Control in Severe Traumatic Injury: a Randomized Controlled Trial
Brief Title: Ketamine for Pain Control After Severe Traumatic Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Thomas Carver, Associate Professor, General Surgery, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO#00037017
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-07

CONDITIONS: Hospital Inpatient Trauma Injury; Pain Management
MeSH Terms: conditions — Agnosia | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine arm (Experimental): Early ketamine infusion therapy at a rate of 3 mcg/kg/min. All ketamine infusions will be calculated based on ideal body weight (IBW), unless actual body weight is less than ideal. Ketamine infusion therapy will be continued for 48 hours. At 2-4 hours post-infusion the patient's pain will be reassessed. If the NPS is more than 5 the infusion will be increased to 5mcg/kg/min. Following each change in the infusion rate the patient's pain will be reassessed at 2-4 hours and adjustments made accordingly. Maximum infusion rate will be set at 9mcg/kg/min. Conversely, The RAAPS team should be notified if neurologic symptoms (hallucinations, delusions, disturbing dreams, vertigo) are developing and, at the discretion of the RAAPS service, a single dose of lorazepam or midazolam may be utilized. The infusion can be decreased from in 2 mcg/kg/min increments if there are symptoms believed to be related to the infusion that do not respond to benzodiazepines.
  Interventions: Drug: Ketamine
- Placebo arm (Placebo Comparator): The 65 patients randomized to the control arm will receive placebo saline solution at a rate equivalent.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Ketamine infusion
  Arms: Ketamine arm
Drug: Placebo — Placebo infusion
  Arms: Placebo arm

SUMMARY:
This study evaluates if the early utilization of ketamine infusion therapy among acutely injured adult trauma hospital inpatients with an ISS >15 will decrease the amount of opioid pain medication used as compared with placebo group. Ketamine infusion therapy initiated within 12 hours of hospital arrival will lead to decreased total opiate consumption (standardized to oral morphine equivalent units) in the first 24 and 48 hours compared to controls.

DETAILED DESCRIPTION:
Traumatically injured hospital inpatients aged 18 - 64 will be enrolled into the study within 24 hours of admission to the hospital. The patients randomized to the experimental arm will receive early ketamine infusion therapy at a rate of 3 mcg/kg/min. All ketamine infusions will be calculated based on ideal body weight (IBW), unless actual body weight is less than ideal. IBW will be calculated for males as 50kg + 2.3*(number of inches above 5 feet) and for women as 45.5kg + 2.3*(number of inches over 5 feet). The 65 patients randomized to the control arm will receive placebo saline solution at a rate equivalent. Time zero will be defined as the time at which the "ketamine / placebo" infusion is begun. For inclusion in the study, initiation of ketamine / placebo infusions must take place within 12 hours of presentation to Froedtert Memorial Lutheran Hospital (FMLH).

Prior to starting the investigational infusion, a single IV push of 50mcg of fentanyl will be administered to any patient with a numeric pain score between 7-10. This is done to achieve more rapid pain control as poor pain control has been shown to lead to higher rates of chronic pain and PTSD.

Patient controlled analgesia will be provided using either morphine or hydromorphone with an initial starting dose of Morphine (1.5mg bolus, 12 min lockout, no continuous rate) or Hydromorphone (0.2mg, 12 min lockout, no continuous rate). Dose or lockout adjustments to the PCA should be done only after first adjusting the Investigational Drug dose. For example, if a patient continues to complain of severe pain (≥6) after 2-4 hours of initiation of the Investigational Drug then the rate of the infusion should be increased (as described below). The adjustments can be initiated by either the RAAPS team or Trauma service. No more than 1 change to PCA or Investigational Drug rate should be performed every 4 hours (ie if PCA was adjusted at midnight, then an adjustment to the Investigational Drug should not be made before 4 am).

At the completion of the 48-hour infusion the inpatient team has the option of transitioning the patient from the PCA to oral pain medications. Additional adjuncts to pain control including epidural or other regional techniques are at the discretion of the primary team but ideally would be delayed until the investigational infusion is completed.

Ketamine infusions will be prepared by the IDS service but will be hung and administered by the inpatient nursing staff. Ketamine infusion therapy will be continued for 48 hours. At 2-4 hours post-infusion the patient's pain will be reassessed. If the NPS is more than 5 the infusion will be increased to 5mcg/kg/min. Following each change in the infusion rate the patient's pain will be reassessed at 2-4 hours and adjustments made accordingly. Maximum infusion rate will be set at 9mcg/kg/min. Conversely, The RAAPS team should be notified if neurologic symptoms (hallucinations, delusions, disturbing dreams, vertigo) are developing and, at the discretion of the RAAPS service, a single dose of lorazepam or midazolam may be utilized. The infusion can be decreased from in 2 mcg/kg/min increments if there are symptoms believed to be related to the infusion that do not respond to benzodiazepines.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64
* ISS >15
* Infusion can be started within 24 hrs of arrival to FMLH (time of injury irrelevant)
* Admitted to Inpatient hospital trauma service (not Ortho/Plastics/Neurosurgery etc)

Exclusion Criteria:

* Age <18 or >64
* History of adverse reaction to ketamine therapy
* Chronic opioid therapy defined as > 3 weeks of >30mg oral morphine equivalents per day
* Current substance abuse with opioids including prescription and/or heroin
* Intubation on arrival or need for urgent intubation on arrival
* GCS <13, significant traumatic brain injury, or suspicion of elevated intracranial pressure resulting in the patient's inability to communicate
* History of psychosis
* Active delirium
* Glaucoma
* Ischemic heart disease defined as active acute coronary syndrome
* Severe, poorly controlled hypertension (SBP >200) on more than two readings
* Aortic Injury requiring HR and BP control
* Concurrent use of monoamine oxidase inhibitors (MAOIs)
* Pregnancy
* Prisoners
* Inability to start investigational drug infusion within 24 hours of arrival

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Cumulative opioid morphine equivalent dose | The first 24 hours
  The cumulative OME will be compared within the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Carver, MD, Principal Investigator — Medical College of WI
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for prevention of post-traumatic stress disorder (PTSD) in individuals experiencing acute traumatic stress symptoms. Cochrane Database Syst Rev. 2024 May 20;5(5):CD013613. doi: 10.1002/14651858.CD013613.pub2. PMID 38767196
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for universal prevention of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2022 Feb 10;2(2):CD013443. doi: 10.1002/14651858.CD013443.pub2. PMID 35141873